CLINICAL TRIAL: NCT04211883
Title: Project ACTIVE: A Randomized Controlled Trial of Personalized and Patient-Centered Preventive Care
Brief Title: Project ACTIVE a Clinical Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-01865
Record Dates: First submitted 2019-12-05; First posted 2019-12-26 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Alcohol Abuse; Obesity
MeSH Terms: conditions — Alcoholism; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active intervention (Experimental): Participants will come to the Project Active clinic and be asked questions about their health history, assist in their health goals, medications will be adjusted, lab work and screening tests will be ordered. At end of each visit, current health recommendations and goals as well as previous health changes will be given after each visit.
  Interventions: Behavioral: ACTIVE intervention
- Standard Clinical Treatment (No Intervention): Participants will continue with their usual clinic care.

INTERVENTIONS:
Behavioral: ACTIVE intervention — The Project ACTIVE intervention was adapted to suit workflow demands of our busy inner-city clinic: (1) identify patients who could most benefit from improvements in adherence to evidence-based preventive care, (2) use a validated mathematical model to quantify and rank the estimated amount of health benefit that would arise from improved adherence to each USPSTF preventive care guideline, (3) communicate this information in a manner informed by risk communication studies relevant to patients from disparate cultural groups and with low literacy and numeracy, (4) engage the patient in a shared decision making process in which the patient identified which preventive health goals aimed to achieve, and (5) set particular action steps for the next visit that were congruent with these goals .
  Arms: Active intervention

SUMMARY:
This is a clinical Randomized Controlled Trial where the study personnel will run a personalized prevention clinic with patients in attempts to improve their preventive health outcomes and compare their health outcomes with a matched control sample of patients who do not receive the clinical intervention.

DETAILED DESCRIPTION:
The Project ACTIVE intervention was constructed around the following framework, and then adapted to suit workflow demands of a busy inner-city clinic: (1) identify patients who could most benefit from improvements in adherence to evidence-based preventive care, (2) use a validated mathematical model that was published in Annals of Internal Medicine to quantify and rank the estimated amount of health benefit that would arise from improved adherence to each USPSTF preventive care guideline, with estimates personalized based on that patient's risk factors and medical history, (3) communicate this information in a manner informed by risk communication studies relevant to patients from disparate cultural groups and with low literacy and numeracy, (4) engage the patient in a shared decision making process in which the patient identified which preventive health goals patient aimed to achieve, and (5) set particular action steps for the next visit that were congruent with these goals. The program supplements rather than substitutes for normally scheduled primary care visits, and is coordinated with these visits whenever possible.

ELIGIBILITY:
Inclusion Criteria:

* Non-elderly non-pregnant adults already in care at Bellevue Ambulatory adult care clinic
* Subjects with at least one of twelve unfulfilled clinical management goals from USPSTF Grade A and B recommendations
* English or Spanish speaking
* Capable of understanding informed consent.

Exclusion Criteria:

* Age >65
* Pregnant
* Dominant comorbidity (one that disproportionately impacts care plans and/or life expectancy).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Change in number of unfulfilled health care goals resulting from USPSTF recommendations over the course of one year | Visits 4 weeks, 8 weeks, 12 weeks, 16 weeks, 28 weeks, 40 weeks
  At follow up visits the patient's data and goal achievement (or lack thereof) is updated into the model along with their new vital signs, lab work, screenings, and medication changes that occurred since their last visit, to enable the model to yield updated results. If the patient has made improvements to their health since the last visit, this is depicted graphically on an updated summary chart, demonstrating what they accomplished since their previous visit.

SECONDARY OUTCOMES:
Change in life expectancy including smoking, hypertension, hyperlipidemia, quality of life. | Visits 4 weeks, 8 weeks, 12 weeks, 16 weeks, 28 weeks, 40 weeks
  Subject will meet with the health coach, who helps the patients meet their health goals in practical ways by setting corresponding behavioral goals. Motivational interviewing techniques are again used, and the patient ends the visit with clear behavioral goals they have created for the next visit. The goals are written out at the bottom of the patient's visual graph depicting the possible health gain. Educational materials and resources are also given to the patient depending on their specific needs, such as food logs to record their diets, lists of local gyms near their residence and lists of healthy foods to buy when grocery shopping. At the end of the visit, a copy of the patient's visual graph with their specific goals are left in the clinic mailbox of their primary care clinician, and notes are documented by the nurse practitioner and the health coach into the electronic medical record system.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Braithwaite, MD, Principal Investigator — NYU Langone

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.Upon reasonable request Requests should be directed to melanie.applegate@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Applegate M, Scott E, Taksler GB, Sanchez M, Duong N, Mark L, Caniglia E, Wallach A, Braithwaite RS. Project ACTIVE: a Randomized Controlled Trial of Personalized and Patient-Centered Preventive Care in an Urban Safety-Net Setting. J Gen Intern Med. 2021 Mar;36(3):606-613. doi: 10.1007/s11606-020-06359-z. Epub 2021 Jan 14. PMID 33443695